CLINICAL TRIAL: NCT01559766
Title: Estimating Dietary Vitamin A Requirement in Chinese Children by Stable-isotope Dilution Technique
Brief Title: Dietary Vitamin A Requirement in Chinese Children and the New Technology of Dietary Assessment
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: ShiYan Centre for Disease Control and Prevention (Unknown); Tufts Medical Center (Other)
Responsible Party: Principal Investigator, Xiufa Sun, Professor, Huazhong University of Science and Technology
Other Study IDs: No.2008BAI58B03
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Vitamin A Deficiency
Keywords: Vitamin A; Dietary requirement; Dietary records; Deuterated retinol dilution technique; Chinese children; Dietary intake of vitamin A; Vitamin A liver reserves
MeSH Terms: conditions — Vitamin A Deficiency

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 4-6 years old group
- 7-9 years old group

SUMMARY:
Vitamin A deficiency remains a major public health problem in developing country worldwide. Young Children are considered to be at greatest risk of deficiency. However, there is little information on the vitamin A requirement of Chinese children. In the present study, about 400 children aged between 4 and 9 years old in a kindergarten and an elementary school of Shiyan City were screened before admission by questionnaire and anthropometric measurement. The vitamin A status of children was assessed by serum vitamin A level, relative dosage reaction and stable-isotope dilution technique. At the same time, their dietary vitamin A intakes were estimated by weighted-food dietary survey. The dietary vitamin A requirement in young children was determined on the basis of dietary vitamin A intakes in Children with adequate vitamin A level.

ELIGIBILITY:
Inclusion Criteria:

* well-nourished children with normal serum retinol(>=1.40umol/L)

Exclusion Criteria:

* ongoing or previous illnesses,
* having taken nutritional supplements within 3 months,
* positive results in the fat absorption test or parasite test,
* increased level of CRP (> 8 mg/L), or
* lower serum level of retinol (< 1.40 umol/L)

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study was carried out in a kindergarten and an elementary school in Shiyan city, Hubei province of China. Initially, 201 kindergarten children (4-6 years old) and 202 grade children (7-9 years old) were subjected to a questionnaire survey on personal information, medical history and dietary habits including dietary supplements.ongoing or previous illnesses, having taken nutritional supplements within 3 months, positive results in the fat absorption test or parasite test, increased level of CRP (> 8 mg/L), or lower serum level of retinol (<1.40 umol/L), and higher ratio in relative dosage reaction test(>20%) .After the screening, 123 children were selected and completed the study, but 60 subjects were randomly selected for the DRD test to evaluate liver vitamin A storage.
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiufa Sun, BS, Principal Investigator — Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Shiyan Centre for Disease Control and Prevention, Shiyan, Hubei, China